CLINICAL TRIAL: NCT02227836
Title: Efficacy of Allergy Patch Testing in Directed Dietary Therapy of Eosinophilic Esophagitis: A Pilot Study
Brief Title: Value of Patch Testing in Direct Diet Therapy for Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-002050; UL1TR000135 (NIH)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: Allergy Patch testing; Eosinophilic Esophagitis; EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Patch Tests; Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allergy Patch Testing APT (Experimental): Patient will undergo APT testing per the following protocol:
  * 2g of dry foods will be placed in 2ml of isotonic saline solution. The mixtures will then be placed in aluminum cups (ie Finn chambers) measuring 6 or 12 mm in diameter and adhered to the patient's back.
  * Foods to be included will be milk, wheat, egg, soy, peanut, tree nut, fish, shellfish, beef, corn, chicken, potato, pork, legumes, barley, rye, tomato, rice, fruits
  * The patches will be removed at 48 hours, and results read at 72 and 120 hours after application
  * Reactions will be classified as negative, + (erythema and scattered papules), ++ (erythema and papules), and +++ (erythema and vesicles).
  Interventions: Device: Allergy Patch Testing

INTERVENTIONS:
Device: Allergy Patch Testing
  Other Names: APT; Patch testing; Allergy testing

SUMMARY:
This study is being done to see if allergy patch testing (APT) can help predict effective dietary therapy in patients with eosinophilic esophagitis.

DETAILED DESCRIPTION:
Patients are referred to Mayo Clinic Rochester with an establish diagnosis of EoE and are nonresponsive to proton pump inhibitor (PPI) medical therapy. Eligible patients will then meet with one of three investigators complete the Mayo Dysphagia Questionaire-30 Day (MDQ-30) following which a standardized Allergy Patch testing (APT) will be conducted. Thereafter, a standard clinically indicated Six Food Elimination Diet treatment completed. Patients will follow up with one of three investigators following the elimination diet who will be blinded to the results of the APT. During this visit responders and nonresponders will be identified and nonresponders will complete a directed elimination diet based on APT results.

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-90
* Patients with EoE, defined as dysphagia with histologic finding of greater than or equal to 15 eosinophils per high powered field (eos per HPF) on index esophageal biopsy
* Persistent symptoms and/or greater than or equal to 10 eos per HPF on esophageal biopsy after at least 8 weeks of twice daily PPI therapy

Exclusion criteria:

* Patients with conditions known to be associated with esophageal eosinophilia, including Crohn's disease, Churg-Strauss, achalasia, and hypereosinophilic syndrome
* Topical swallowed steroids within 8 weeks of study enrollment
* Dermatologic conditions precluding application of Finn chambers to the skin for APT
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eckmann JD, Ravi K, Katzka DA, Davis DR, See JA, Geno DR, Kryzer LA, Alexander JA. Efficacy of Atopy Patch Testing in Directed Dietary Therapy of Eosinophilic Esophagitis: A Pilot Study. Dig Dis Sci. 2018 Mar;63(3):694-702. doi: 10.1007/s10620-018-4928-4. Epub 2018 Jan 18. PMID 29349695
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Allergy Patch Testing APT: Patient will undergo Atopy Patch Testing (APT) per the following protocol:
  * 2g of dry foods will be placed in 2ml of isotonic saline solution. The mixtures will then be placed in aluminum cups (ie Finn chambers) measuring 6 or 12 mm in diameter and adhered to the patient's back.
  * Foods to be included will be milk, wheat, egg, soy, peanut, tree nut, fish, shellfish, beef, corn, chicken, potato, pork, legumes, barley, rye, tomato, rice, fruits
  * The patches will be removed at 48 hours, and results read at 72 and 120 hours after application.
  * Reactions will be classified as negative, + (erythema and scattered papules), ++ (erythema and papules), and +++ (erythema and vesicles).
Period: Overall Study
Arm/Group | Allergy Patch Testing APT
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Allergy Patch Testing APT: Patient will undergo APT testing per the following protocol:
  * 2g of dry foods will be placed in 2ml of isotonic saline solution. The mixtures will then be placed in aluminum cups (ie Finn chambers) measuring 6 or 12 mm in diameter and adhered to the patient's back.
  * Foods to be included will be milk, wheat, egg, soy, peanut, tree nut, fish, shellfish, beef, corn, chicken, potato, pork, legumes, barley, rye, tomato, rice, fruits
  * The patches will be removed at 48 hours, and results read at 72 and 120 hours after application.
  * Reactions will be classified as negative, + (erythema and scattered papules), ++ (erythema and papules), and +++ (erythema and vesicles).
Arm/Group | Allergy Patch Testing APT
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Allergic history [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Patch Testing
Description: Sensitivity of the patch test will be defined by the number of subjects with total positive APT reactions correlated to histologic findings
Time Frame: up to 120 hours after application of patch test
Measure: Count of Participants; unit: Participants
Groups:
- Allergy Patch Testing APT: Patient will undergo APT testing per the following protocol:
  * 2g of dry foods will be placed in 2ml of isotonic saline solution. The mixtures will then be placed in aluminum cups (ie Finn chambers) measuring 6 or 12 mm in diameter and adhered to the patient's back.
  * Foods to be included will be milk, wheat, egg, soy, peanut, tree nut, fish, shellfish, beef, corn, chicken, potato, pork, legumes, barley, rye, tomato, rice, fruits
  * The patches will be removed at 48 hours, and results read at 72 hours after application.
  * Reactions will be classified as negative, + (erythema and scattered papules), ++ (erythema and papules), and +++ (erythema and vesicles).
Arm/Group | Allergy Patch Testing APT
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: Data were collected from baseline until 2 weeks after completion of the final study visit for each subject.
Arm/Group | Allergy Patch Testing APT
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT02227836/Prot_SAP_000.pdf